CLINICAL TRIAL: NCT00322543
Title: Reduced Anti-Platelet Therapy With Pimecrolimus Drug Eluting Stent (RAPID) A Multi-Center Study of the Pimecrolimus-Eluting Cobalt Chromium Coronary Stent System (Corio™) in Patients With De Novo Lesions of the Native Coronary Arteries
Brief Title: Reduced Anti-Platelet Therapy With Pimecrolimus Drug Eluting Stent (RAPID)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Conor Medsystems (Industry)
Responsible Party: Alexandre Abizaid, MD, Institute Dante Pazzanese of Cardiology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAPID (Genesis) Registry CP-02
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-09

CONDITIONS: Coronary Disease
Keywords: Percutaneous coronary intervention (PCI); Drug eluting stent (DES)
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug eluting stent (Experimental): Corio™ Pimecrolimus-eluting stent
  Interventions: Device: Corio™ Pimecrolimus-eluting stent

INTERVENTIONS:
Device: Corio™ Pimecrolimus-eluting stent

SUMMARY:
Non-randomized, single arm, multi-center, clinical trial evaluating the Corio™ pimecrolimus-eluting stent with reduced anti-platelet therapy in patients with de novo lesions of the native coronary arteries.

DETAILED DESCRIPTION:
The registry is designed to evaluate 6-month in-stent late lumen loss in patients receiving the Corio™ drug-eluting stent.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Eligible for percutaneous coronary intervention (PCI).
2. Documented stable or unstable angina pectoris
3. Left ventricular ejection fraction (LVEF) ≥25%
4. Acceptable candidate for coronary artery bypass graft surgery (CABG).
5. Target Lesion < 25 mm in length with RVD of 2.5 to 3.5 mm with visually estimated stenosis of >= 50 and < 100 %.

Exclusion Criteria:

General Exclusion Criteria

1. Known sensitivity to pimecrolimus, the polymer (PLGA) or cobalt chromium.
2. Planned treatment with any other PCI device in the target vessel(s).
3. MI within 72 hours prior to the index procedure
4. The patient is in cardiogenic shock.
5. Cerebrovascular Accident (CVA) within the past 6 months.
6. Acute or chronic renal dysfunction
7. Contraindication to ASA or to clopidogrel.
8. Thrombocytopenia
9. Active gastrointestinal (GI) bleeding within the past 3 months.
10. Any prior true anaphylactiod reaction to contrast agents
11. Patient is currently taking chronic systemic steroid therapy or systemic immunosuppressant therapy or topical pimecrolimus.
12. Female of childbearing potential.
13. Life expectancy of less than 24 months due to other medical conditions.
14. Co-morbid condition(s)
15. Currently participating in another investigational drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-05; Primary Completion 2006-11 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Angiographic endpoint of in-stent late lumen loss at 6 months | 6 months

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) defined as an adjudicated composite of clinically driven target vessel revascularization, new myocardial infarction (MI) or cardiac death at 30 days, 6 months, 12 months and 2 years; | 30 days, 6 months, 12 months and 2 years
Device, Lesion and Procedural Success; Coronary angiography at 6 months; IVUS measurements in IVUS cohort at 6 months. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Abizaid, M.D., Principal Investigator — Institute Dante Pazzanese of Cardiology
Locations (1):
- Institute Dante Pazzanese of Cardiology, São Paulo, São Paulo, Brazil